CLINICAL TRIAL: NCT02699970
Title: Instrument Precision Study for Validation of Philips Dx
Status: Completed | Type: Observational
Sponsor: Philips Digital & Computational Pathology (Industry)
Responsible Party: Sponsor
Other Study IDs: DPS-CT-0009
Record Dates: First submitted 2016-03-01; First posted 2016-03-07 (Estimated); Results first posted 2019-11-01 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Pathology

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Selected features: No intervention is administered to the selected features. They only need to be observed by the pathologist.
  The features are part of tissue that is present on a slide. This slide is fully scanned and the digital image is than viewed by the pathologist who indicates if he can see the feature. By repeating the scan three times and having the pathologist view three times, the consistency of the feedback can be monitored. The consistency is a measure on how repeatable and reproducible the scanner is. To be very clear: the scanner does not do anything to the tissue. It only takes a digital 'photo' of the tissue. It is no treatment or intervention. It just takes a picture.

SUMMARY:
The objective of this study is to evaluate precision of the Philips Dx system.

DETAILED DESCRIPTION:
Slides were selected that contained clinically relevant histopathologic "features" that are generally encountered on surgical pathology slides. Twenty-one features, each selected from three different organs, were to be included to ensure that multiple tissue types were investigated. The study feature(s) as selected on each slide was defined as the "selected feature". In total 420 selected features were acquired and the slides holding these features composed the "slide set". The slideset consisted of 399 slides from 399 different participants.

1. Intra-system study. The full slide set was then divided over three subsets. Each subset was then scanned three times on one systems, with each subset being scanned on a different scanner. This means that each feature was scanned three times. Each of three pathologists read all three scans of the entire slide set. Intra-system precision was thereby determined.
2. Inter-system study. The full slide set was then scanned three times, each time on a different system, meaning that each feature was scanned three times. Each of three pathologists (different pathologists the ones used in the intra-system study) read all three scans of the entire slide set. Inter-system precision was thereby determined.

ELIGIBILITY:
Inclusion Criteria:

* Left-over specimens from subjects who already received their diagnosis and have received their treatment in accordance with the standard of care
* H&E glass coverslipped slides with human tissue obtained via surgical pathology
* Selected slides fulfill the quality checks according to the Instructions for Use (lfU)
* Selected slides must be between 1-5 years since accessioning
* Selected slides and FOVs must contain a study feature that is: In it's natural environment (on slide and FOV); Readily observable (on slide and FOV); Not equivocal (on slide and FOV).

Exclusion Criteria:

* Selected slides contain indelible markings
* Selected slides contain damaged tissue
* More than one slide was selected for a patient (only one slide may be enrolled per patient).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cases will be selected from the LIS in consecutive order. Cases will be selected per feature and per organ. From these cases, slides will be selected containing the pre-specified study feature.
Sampling Method: Non-Probability Sample
Enrollment: 399 (Actual)
Dates: Start 2016-02; Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mischa Nelis, Study Director — Philips DPS
Locations (1):
- MGH, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started enrollment in February 2016 and enrollment was completed in April 2016. The full set of 420 features were used for the intra-system study as well as for the inter-system sub-study.
Pre-assignment Details: Features were evenly distributed over three magnifications (10x, 20x or 40x). 21 different feature types were included. Each feature type was divided over three organs.
Units Other Than Participants: feature
Groups:
- Precision: Intra-system: At one study site the slides with selected features were evenly distributed over three different systems. Each slide was scanned three times on the same system. All scans were read by all three pathologists.
  Inter-system: At one study site the full set of slides with selected features was scanned once on three different scanners. All three pathologists read all scans.
Period: Overall Study
Arm/Group | Precision
Started | 399; 420 feature
Intra-system | 399; 420 feature
Inter-system | 399; 420 feature
Completed | 399; 420 feature
Not Completed | 0; 0 feature

BASELINE CHARACTERISTICS:
Population: Features for intra-system sub-study were also used for inter-system sub-study. Baseline characteristics were not considered relevant and therefore not collected in this study.
Units Other Than Participants: features
Arm/Group | Precision
Number analyzed (Participants) | 399
Number analyzed (features) | 420
Age, Categorical [Count of Participants; unit: Participants] — Population: Data were considered not relevant and therefore were not collected
  Participants
    number analyzed (Participants) | 0
Sex: Female, Male [Count of Units; unit: features] — Population: Data were considered not relevant and therefore were not collected
Region of Enrollment [Number; unit: Study features]
  United States | 420

OUTCOME MEASURES:

1. Primary Outcome: Agreement Rate
Description: The agreement rate between reads calculated over all selected features and pathologists. Readings were considered in agreement when the selected feature was indicated as 'present' or 'absent' in both readings.
Time Frame: 2 months
Population: For the intra-system sub-study 2 cases were not analyzed for possible reading bias due to an error in the EDC system.
  For the inter-system sub-study 3 cases were not analyzed for different reasons such as possible reading bias due to an error in the EDC system (2) and a short washout period (1).
Measure: Mean (95% Confidence Interval); unit: percentage of agreement
Units Other Than Participants: features
Groups:
- Intra-system Sub-study: At one study site the slides with selected features were evenly distributed over three different systems. Each slide was scanned three times on the same system. All scans were read by all three pathologists.
- Inter-system Sub-study: At one study site the full set of slides with selected features was scanned once on three different scanners. All three pathologists read all scans.
Arm/Group | Intra-system Sub-study | Inter-system Sub-study
Number analyzed (Participants) | 397 | 396
Number analyzed (features) | 418 | 417
percentage of agreement | 92.0 [90.57 to 93.29] | 93.8 [92.56 to 94.98]

ADVERSE EVENTS:
Time Frame: From study start to study closure (8 months)
Groups:
- Precision: Intra-system sub-study: At one study site the slides with selected features were evenly distributed over three different systems. Each slide was scanned three times on the same system. All scans were read by all three pathologists.
  Inter-system sub-study: At one study site the full set of slides with selected features was scanned once on three different scanners. All three pathologists read all scans.
Arm/Group | Precision
All-Cause Mortality (participants affected / at risk) | 0/399
Serious Adverse Events (participants affected / at risk) | 0/399
Other Adverse Events (participants affected / at risk) | 0/399

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less